CLINICAL TRIAL: NCT01000584
Title: PCIRN Evaluation of Pandemic H1N12009 Influenza Vaccine in Adults, Including Randomized Comparison of Concurrent or Delayed Seasonal Influenza Vaccination
Brief Title: Rapid Evaluation of Pandemic H1N1 Influenza Vaccine in Adults Receiving Seasonal Influenza Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: David Scheifele (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, David Scheifele, Director Vaccine Evaluation Center, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H09-02811
Record Dates: First submitted 2009-10-21; First posted 2009-10-23 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Influenza; H1N1 2009 Influenza
Keywords: vaccine; H1N1; influenza; H1N1 influenza vaccine; influenza vaccine; seasonal Influenza
MeSH Terms: conditions — Influenza, Human | interventions — arepanrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Group A: One dose of the licensed H1N1 vaccine and one dose of the seasonal influenza vaccine given concurrently
  Interventions: Biological: Arepanrix, Vaxigrip 2009/2010
- 2 (Other): Group B: One dose of seasonal influenza vaccine given 3 weeks after administration of one dose of the licensed H1N1 vaccine
  Interventions: Biological: Arepanrix, Vaxigrip 2009/2010

INTERVENTIONS:
Biological: Arepanrix, Vaxigrip 2009/2010 — Group A: Single dose of Arepanrix and single dose of Vaxigrip 2009/2010 given concurrently
  Arms: 1
Biological: Arepanrix, Vaxigrip 2009/2010 — Group B: Single dose of Vaxigrip 2009/2010 given 3 weeks after single dose of Arepanrix
  Arms: 2

SUMMARY:
The purpose of this study is to assess the safety and effectiveness (immune response) to a licensed H1N12009 influenza vaccine in adults when given at the same time or prior to the seasonal influenza vaccine. The study will enroll 300 adults (ages 20-59 years). Participants will be randomized into 2 groups. One group will receive one dose of a licensed H1N1 vaccine and one dose of the seasonal influenza vaccine at the same time; the second group will receive the seasonal influenza vaccine 3 weeks after receiving the licensed H1N12009 influenza vaccine. Study procedures include: medical history, blood samples and completing a memory aid. Participants will be involved in study related procedures for approximately 3-6 weeks depending upon the group assignment.

DETAILED DESCRIPTION:
The objectives of this study are two-fold:

1. To evaluate the safety and immunogenicity of H1N12009 influenza vaccine in a convenience sample of adults, soon after the pandemic vaccine becomes available so as to inform the subsequent use of vaccine in public programs.
2. To evaluate the compatibility of co-administered H1N12009 pandemic vaccine and seasonal TIV vaccine in the same group of subjects, as the option of co-administration would be useful for public programs.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adults 20-59 years of age

Exclusion Criteria:

* Allergies to eggs, thimerosal, gentamicin sulphate, neomycin
* Life-threatening reaction to previous Flu vaccine
* Bleeding disorder
* Pregnancy
* Receipt of blood or blood products in past 3 months
* Chronic illness
* Compromised immune system
* Previous lab-confirmed H1N12009 infection
* Receipt of H1N12009 vaccine
* Receipt of Seasonal Influenza vaccine since March 2009

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 309 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs) for days 0-6 after each vaccination | Day 7 and Day 21 post vaccination
Occurrence of serious adverse events (SAEs) and other significant health events up to 21 days after each vaccination | Day 7 and Day 21 post vaccination

SECONDARY OUTCOMES:
Immunogenicity: Comparison of baseline and post-immunization antibody titres | Day 21 post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: David Scheifele, MD, Principal Investigator — University of British Columbia; Allison McGeer, MD, Study Director — University of Toronto, Mt Sinai Hospital; Mark Loeb, MD, Study Director — McMaster University; Ian Gemmill, MD, Study Director — Kingston, Frontenac, Lanark Health Unit; Marc Dionne, MD, Study Director — Institut national de sante publique du Quebec
Locations (4):
- Canada (4):
  - McMaster University, Hamilton, Ontario
  - Kingston, Frontenac, Lanark Health Unit, Kingston, Ontario
  - University of Toronto, Mt Sinai Hospital, Toronto, Ontario
  - Institut national de sante publique du Quebec, Québec, Quebec

REFERENCES:
- [Derived] Scheifele DW, Ward BJ, Dionne M, Vanderkooi OG, Loeb M, Coleman BL, Li Y; PHAC/CIHR Influenza Research Network (PCIRN). Compatibility of ASO3-adjuvanted H1N1pdm09 and seasonal trivalent influenza vaccines in adults: results of a randomized, controlled trial. Vaccine. 2012 Jul 6;30(32):4728-32. doi: 10.1016/j.vaccine.2012.05.029. Epub 2012 May 28. PMID 22652402